CLINICAL TRIAL: NCT04533139
Title: Effect of Annual Influenza Immunization on Antibody Response in Lung Transplant Patients
Brief Title: Influenza Vaccine in Lung Transplant Patients - Antibody
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2004-0240b; A561000 (Other: UW Madison); PHARM/PHARMACY/PHARMACY (Other: UW Madison)
Record Dates: First submitted 2020-08-25; First posted 2020-08-31 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Influenza
Keywords: Pre or post-lung transplant; Healthy
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vaccine, pre-transplant: cohort consists of individuals waiting for lung transplantation. Inactivated influenza vaccine will be administered intramuscularly annually.
  Interventions: Drug: Influenza vaccine
- Vaccine, post-transplant: Cohort consist of individuals who have received lung transplants Inactivated influenza vaccine will be administered intramuscularly annually.
  Interventions: Drug: Influenza vaccine
- Vaccine, not receiving transplant: Cohort consists of healthy individuals who received the influenza vaccine Inactivated influenza vaccine will be administered intramuscularly annually.
  Interventions: Drug: Influenza vaccine

INTERVENTIONS:
Drug: Influenza vaccine — influenza vaccine 0.5 ml intramuscularly each season
  2004-2005 season antigens: A/New Caledonia/20/99(H1N1)-like, A/Wyoming/3/2003(H3N2), and B/Shanghai/361/2002-like antigens
  2005-2006 season antigens: A/New Caledonia/ 20/00(H1N1)-like, A/California/7/2004 (H3N2)-like, and B/Shanghai/361/2002-like antigens

SUMMARY:
This is a sub-study of a 5-year study designed to investigate how antibody and T cell responses following influenza vaccine compare among lung transplant patients, patients waiting for lung transplantation, and healthy individuals.

This prospective, parallel study was done to investigate the responses to influenza vaccine in consecutive years.

DETAILED DESCRIPTION:
Lung transplant patients may be at an incrementally higher risk of influenza infection than other transplant patients. Factors that predispose them to respiratory infection include high degree of immunosuppression, altered mucociliary clearance, repeated airway instrumentation, bronchial anastomotic obstruction, disruption of lymphatic drainage, and the exposure of the transplanted organ to the environment.

The influenza vaccine used for those at high risk for influenza morbidity and mortality is an inactivated trivalent preparation. Influenza vaccine contains 2 type A viruses and 1 type B virus. The vaccine is reformulated each year based on the viruses expected to circulate during the upcoming season. A protective antibody response to influenza vaccine is considered an antibody titer of at least 1:40. Seroconversion following influenza immunization implies at least a 4-fold increase in antibody concentrations. Although these indicators of a positive response to influenza immunization have significant overlap, they are not exactly the same. One must consider that a person may have antibodies before immunization because of previous exposure to a vaccine virus or an antigenically similar influenza strain.

Seroconversion rates following influenza vaccination are lower in lung transplant patients than in healthy persons. Clearly, immunization elicits an antibody response in this population, but the response is not as vigorous as in immunocompetent persons. It has been demonstrated that only the B/HongKong virus was associated with a lower seroconversion rate, and this virus was the only one to change from the previous year's vaccine. Seroconversion rates decrease with subsequent exposure to the same influenza vaccine viruses, but seroprotection rates remain the same. It is conceivable that the seroconversion response is more affected by immunosuppression than is the seroprotection response. Stated another way, the ability to mount a high spike in antibody production is hindered. It is difficult to fully ascertain the exact degree of immune impairment in lung transplant recipients because both studies investigating influenza vaccine response used healthy persons as the comparison group. Healthy persons may have less experience with influenza vaccine than do persons with severe respiratory conditions. An immunologically naive host is more likely to mount the large change in antibody concentration and increase the likelihood of seroconversion. Therefore, patients waiting for lung transplantation were used as a comparison group.

This prospective, parallel study was done to investigate the responses to influenza vaccine in consecutive years. All participants had a blood sample taken for measurement of influenza antibody titers before receiving the influenza vaccine. Subsequently, the 2004-2005-A/New Caledonia/20/99(H1N1)-like, A/Wyoming/3/2003(H3N2), and B/Shanghai/361/2002-like antigens-and/or 2005-2006-A/New Caledonia/ 20/00(H1N1)-like, A/California/7/2004 (H3N2)-like, and B/Shanghai/361/2002-like antigens-influenza vaccine was administered intramuscularly. Serum was stored at -80°C until the day of analysis. A second blood sample was obtained 2 to 4 weeks later to measure antibody response.

[This substudy that was originally registered to NCT00205270 and subsequently registered to its own NCT number for the purpose of clarity in linked results]

ELIGIBILITY:
Inclusion Criteria:

* Receiving care pre- or post-lung transplant at University of Wisconsin Hospital
* Healthy adult

Exclusion Criteria:

* Allergy to eggs
* Moderate to severe febrile illness
* Active treatment for acute rejection
* Received season's influenza vaccine prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy adults, or patients receiving care pre- or post-lung transplant at University of Wisconsin Hospital
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2004-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Log-transformed change in Antibody Responses | baseline, 2-4 weeks post-vaccination (2004-2005 season), up to 1 year, up to 1 year and 4 weeks (2005-2006 season)
  Influenza antibody concentrations are measured by HIA in samples taken before immunization and 2 to 4 weeks later. Antibody response is the difference in serum concentrations from before and 2 to 4 weeks after vaccination. Antibody concentrations were compared between seasons by using a Wilcoxon rank sum test.

SECONDARY OUTCOMES:
Incidence of Seroconversion | 2-4 weeks post-vaccination (2004-2005 season), up to 1 year and 4 weeks (post-vaccination 2005-2006 season)
  Seroconversion was defined as more than a 4-fold increase in serum hemagglutination units (HAU).
Incidence of Seroprotection | baseline, 2-4 weeks post-vaccination (2004-2005 season), up to 1 year, up to 1 year and 4 weeks (2005-2006 season)
  Seroprotection was defined as an antibody concentration of 40 HAU or greater.
Correlation of Time Since Transplantation to Antibody Response in Lung Transplant Patients | 2-4 weeks post-vaccination (2004-2005 season), up to 1 year and 4 weeks (post-vaccination 2005-2006 season)
  Time since transplant was correlated to antibody responses in the transplant subjects by using a Spearman correlation coefficient to determine the influence of chronic immunosuppression on immune responses. Statistical significance was defined as P less than .05.

CONTACTS AND LOCATIONS:
Overall Officials: Mary S Hayney, PharmD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dopp JM, Wiegert NA, Moran JJ, Francois ML, Radford KL, Thomas H, Love RB, Hayney MS. Effect of annual influenza immunization on antibody response in lung transplant patients. Prog Transplant. 2009 Jun;19(2):153-9. doi: 10.1177/152692480901900209. PMID 19588665